CLINICAL TRIAL: NCT04505267
Title: Phase I Study of Reirradiation With NBTXR3 for Inoperable Locoregional Recurrent Non-Small Cell Lung Cancer (NSCLC)
Brief Title: NBTXR3 and Radiation Therapy for the Treatment of Inoperable Recurrent Non-small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0123; NCI-2020-04580 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0123 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2020-07-14; First posted 2020-08-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Recurrent Lung Non-Small Cell Carcinoma; Stage I Lung Cancer AJCC v8; Stage IA1 Lung Cancer AJCC v8; Stage IA2 Lung Cancer AJCC v8; Stage IA3 Lung Cancer AJCC v8; Stage IB Lung Cancer AJCC v8; Stage II Lung Cancer AJCC v8; Stage IIA Lung Cancer AJCC v8; Stage IIB Lung Cancer AJCC v8; Stage III Lung Cancer AJCC v8; Stage IIIA Lung Cancer AJCC v8; Stage IIIB Lung Cancer AJCC v8; Stage IIIC Lung Cancer AJCC v8; Unresectable Lung Non-Small Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (NBTXR3, RT) (Experimental): Patients receive NBTXR3 IT or intranodally on day 1. Within 15 days, patients undergo RT 5 times weekly (Monday-Friday) over 3 weeks for a total of 10-15 fractions.
  Interventions: Other: Hafnium Oxide-containing Nanoparticles NBTXR3; Radiation: Radiation Therapy

INTERVENTIONS:
Other: Hafnium Oxide-containing Nanoparticles NBTXR3 — Given IT or intranodally
  Other Names: NBTXR3
Radiation: Radiation Therapy — Undergo RT
  Other Names: Cancer Radiotherapy; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation

SUMMARY:
This phase I trial investigates the best dose and side effects of NBTXR3 when given together with radiation therapy for the treatment of non-small cell lung cancer that cannot be treated by surgery (inoperable) and has come back (recurrent). NBTXR3 is a radio-enhancer designed to increase the radiotherapy energy dose deposition inside tumor cells. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. Giving NBTXR3 and radiation therapy may increase radiation-dependent tumor cell killing without increasing the radiation exposure of healthy surrounding tissues.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the safety of 45 Gy in 15 fractions in patients with inoperable, locoregional recurrent NSCLC, previously treated with definitive radiation therapy.

II. To determine the recommended phase II dose (RP2D) of NBTXR3 activated by radiotherapy in patients with inoperable, locoregional recurrent NSCLC, previously treated with definitive radiation therapy.

SECONDARY OBJECTIVES:

I. To evaluate the safety and feasibility of reirradiation with NBTXR3 in patients with inoperable, locoregionally recurrent NSCLC.

II. To evaluate the anti-tumor response of reirradiation with NBTXR3 in patients with inoperable, locoregionally recurrent NSCLC.

III. To evaluate time-to-event outcomes after reirradiation with NBTXR3 in patients with inoperable, locoregionally recurrent NSCLC

EXPLORATORY OBJECTIVE:

I. To assess biomarkers of response in patients treated with NBTXR3/radiation therapy (RT).

OUTLINE: This is a dose-escalation and dose-expansion study of NBTXR3.

Patients receive NBTXR3 intratumorally (IT) or intranodally on day 1. Within 15 days, patients undergo RT 5 times weekly (Monday-Friday) over 3 weeks for a total of 10-15 fractions.

After completion of study treatment, patients are followed up every 3 months for 2 years, then every 6 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy proven locoregionally recurrent NSCLC after prior definitive radiation therapy, or patients that have imaging characteristics highly suggestive of recurrence but no pathologic or cytologic diagnosis. Pathologic diagnosis will be confirmed during the procedure to inject NBTXR3, prior to injecting the drug. If pathologic diagnosis cannot be established, the procedure will be aborted and the patient will be considered a screening failure. For stage IV patients, oligometastatic disease should be confirmed at screening. Oligometastatic disease is defined as ≤ 3 cancer lesions, not including the primary tumor.
2. Participant deemed medically inoperable by the investigator or treating physician.
3. Overlap between recurrent disease in need of treatment and prior radiation treatment field as determined by treating Radiation Oncologist.

   1. As a general reference, recurrent disease within 50% isodose line of prior radiation treatment field would be considered significant.
   2. Radiation treatment received more than 6 months prior to enrollment.
4. Amenable to undergo bronchoscopic (EBUS, CBCT) or CT-guided injection of NBTXR3 as per investigator or treating physician.

   1. Up to 4 lung lesions may be injected with NBTXR3, including the primary tumor, involved lymph node(s), and/or metastatic lesion(s).
   2. At least 1 injected lesion should be located within a reirradiation field.
   3. All injected lesions must be radiated.
5. The target lesion(s) should be measurable on cross sectional imaging (RECIST 1.1).

   a. Nodal target lesions must be ≥15 mm (short axis) based on CT (slice thickness of 5 mm or less) or MRI.
6. Age ≥ 18 years
7. ECOG Performance Status 0-2
8. For cohort 1, adequate laboratory values to receive radiation as determined by the principal investigator or treating physician.
9. For cohort 2 laboratory values at screening:

   1. Hemoglobin ≥ 8.0 g/dL
   2. Absolute Neutrophil Count (ANC) ≥ 1,500/mm3
   3. Platelet Count ≥ 100,000/mm3
   4. Creatinine ≤ 1.5 x upper limit of normal (ULN)
   5. Calc. Creatinine Clearance ≥ 30 mL/min
   6. Total Bilirubin ≤ 2.0 mg/dL
   7. AST / ALT ≤ 3.0 x upper limit of normal (ULN) or 5.0 x ULN if known liver metastases
   8. Serum albumin ≥ 3.0 g/dL
10. Negative urine or serum pregnancy test ≤ 7 days of NBTXR3 injection in all female of child-bearing potential.
11. Signed informed consent form (ICF) indicating that participant understands the purpose of, and procedures required for, the study and is willing to participate in the study.
12. English speaking or Non-English Speaking subjects

Exclusion Criteria:

1. At screening, past medical history of:

   1. Interstitial lung disease, excluding drug-induced ILD, speficially immunotherapy-induced pneumonitis that has been resolved
   2. Any Grade 4 thoracic radiation related toxicity
   3. Unresolved radiation related

   i. Esophagitis ii. Pneumonitis iii. Bronchopulmonary hemorrhage d. Any Grade i. Esophageal perforation ii. Radiation associated airway necrosis iii. Bronchoesophageal fistula e. Any Grade i. Esophageal perforation ii. Radiation associated airway necrosis iii. Bronchoesophageal fistula iv. Tracheoesophageal fistula v. Spinal cord myelopathy
2. Has received any approved or investigational anti-neoplastic or immunotherapy agent within 2 weeks prior to NBTXR3 injection
3. Use of concurrent systemic therapy (chemotherapy, immunotherapy, targeted therapy) or patient participation on another therapeutic clinical trial.
4. Active malignancy, in addition to locoregionally recurrent NSCLC, with the exception of definitively treated and relapse free within 1 year from diagnosis of non-melanoma skin cancer or cervical cancer in situ; definitively treated non-metastatic prostate cancer; or patients with another primary malignancy who are definitively treated and relapse free with at least 2 years elapsed since the diagnosis of the other primary malignancy.
5. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, renal failure, cardiac arrhythmia, or psychiatric illness that would limit compliance with treatment.
6. Known active, uncontrolled (high viral load) HIV or hepatitis B or hepatitis C infection
7. Female patients who are pregnant or breastfeeding.
8. Women of child-bearing potential and their male partners who are unwilling or unable to use an acceptable method of birth control to avoid pregnancy for the entire study period. Acceptable methods of contraception are those that, alone or in combination, result in a failure rate of < 1% per year when used consistently and correctly.
9. Any condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant (e.g., compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments.
10. Cognitively impaired subjects

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicity (DLT) Cohort 1 | Day 1 to 3 months post radiation therapy (RT)
  Defined as the occurrence and frequency of DLTs by dose level of NBTXR3. Descriptive summary tables will be produced, providing the DLTs by initial planned dose level of NBTXR3, initial planned volume of NBTXR3 to be injected, the injected volume and the RT dose given.
Determination of the Recommended Phase II Dose (RP2D) | 4 weeks post RT
  Will be selected based on isotonic regression. Specifically, the recommended phase II dose (RP2D) will be determined as the dose for which the isotonic estimate of the toxicity rate is closest to the target toxicity rate (30%).
Incidence of dose limiting toxicity (DLT) Cohort 2 | Day 1 to 4 weeks post RT
  Defined as the occurrence and frequency of DLTs by dose level of hafnium oxide-containing nanoparticles NBTXR3 (NBTXR3). Descriptive summary tables will be produced, providing the DLTs by initial planned dose level of NBTXR3, initial planned volume of NBTXR3 to be injected, the injected volume and the RT dose given. Incidence of dose-limiting toxicities (DLTs) for NBTXR3 with RT. The DLT window for cohort 2 (NBTXR3 + RT) is from Day 1 to 4 weeks post RT.
Determination of the maximum tolerated dose (MTD) | 4 weeks post RT
  Determination of the MTD will be selected based on isotonic regression. Specifically, the MTD will be determined as the dose for which the isotonic estimate of the toxicity rate is closest to the target toxicity rate (30%).

SECONDARY OUTCOMES:
Incidence of NBTXR3/RT related late onset toxicities | Up to 5 years
  Defined as any grade >= 3 adverse events (AE) occurring after the end of treatment visit and until end of study (EoS). All AEs will be coded and graded according to National Cancer Institute-Common Terminology Criteria for Adverse Events version (v)5 criteria.
Feasibility of NBTXR3 injection in lung | Up to 5 years
  Feasibility is defined as the ability to do intratumoral and/or intranodal lung injection of NBTXR3.
Feasibility of the regional lymph nodes | Up to 5 years
  Feasibility is defined as the ability to do intratumoral and/or intranodal lung injection of NBTXR3.
Objective response rate (ORR) | Up to 5 years
  Defined as the proportion of participants with either a complete response (CR) or a partial response (PR) (ORR=CR + PR) or stable disease (SD) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 and immune-related (ir)RECIST in the target lesion(s) and overall.
Local disease control rate (LDCR) | At 1 and 2 years
  Defined as the proportion of patients who demonstrate a radiographic response to treatment (RECIST v1.1 and irRECIST). The response to treatment should be a CR, PR and/or SD within the selected target lesion(s). Will be estimated by the Kaplan-Meier method. Median times and 95% confidence intervals will also be estimated.
Local progression free survival (LPFS) | From NBTXR3 injection to local (i.e., within the lungs or regional nodes) disease recurrence, local progression, or death from any cause, assessed up to 5 years
  Will be estimated by the Kaplan-Meier method. Median times and 95% confidence intervals will also be estimated.
Distant progression free survival (DPFS) | From NBTXR3 injection to the radiographic confirmation (RECIST v1.1 and irRECIST) of a new lesion outside the lungs and regional nodes or death from any cause, assessed up to 5 years
  Will be estimated by the Kaplan-Meier method. Median times and 95% confidence intervals will also be estimated.
Progression free survival (PFS) | From NBTXR3 injection to local or recurrence, local progression, distant progression, confirmed radiographically (RECIST v1.1 and irRECIST), or death from any cause, assessed up to 5 years
  Will be estimated by the Kaplan-Meier method. Median times and 95% confidence intervals will also be estimated.
Overall survival (OS) | From NBTXR3 injection to death from any cause or EoS, assessed up to 5 years
  Will be estimated by the Kaplan-Meier method. Median times and 95% confidence intervals will also be estimated.

OTHER OUTCOMES:
Tumor microenvironment | Up to 5 years
  Analyzed using multiplexed immunohistochemistry.
Immune activation | Up to 5 years
  Will be quantified by flow cytometry analysis of T and B cells, peripheral blood mononuclear cells.
Circulating tumor deoxyribonucleic acid (DNA) mutations | Up to 5 years
  Will assess the concordance of circulating tumor DNA mutations to those detected in non-small cell lung cancer (NSCLC) tumor-derived DNA.

CONTACTS AND LOCATIONS:
Overall Officials: Saumil Gandhi, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States